CLINICAL TRIAL: NCT06929026
Title: Retinal Biomarkers in Parkinson´s Disease: Retinal Oximetry, Pattern Electroretinography (PERG), Visual Evoked Potentials (VEP) and Optical Coherence Tomography (OCT)
Brief Title: Retinal Biomarkers in Parkinson´s Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Landspitali University Hospital (Other)
Collaborators: Reykjalundur Rehabilitation (Unknown); University of Iceland (Other)
Responsible Party: Principal Investigator, Thorunn Scheving Eliasdottir, Academic chair, Associate Professor, Landspitali University Hospital
Other Study IDs: VSN-22-129
Record Dates: First submitted 2025-03-31; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Retinal oximetry; Pattern Electroretinography; Visual Evoked Potentials; Optical Coherence Tomography; Oxyhemoglobin saturation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine whether oxygen content of the retinal vessels of the eye may serve as a biomarker in Parkinson´s disease. The main questions it aims to answer are:

1. Is retinal vessel oxyhemoglobin saturation and vessel width altered in people with Parkinson´s disease?
2. Is the thickness of the retinal nerve fiber layer altered in people with Parkinson´s disease?
3. Is the response of ganglion cells of the inner retina and the visual cortex altered in people with Parkinson´s disease?

The study procedure is threefold. The participants will:

A. Sit in front of a screen and focus on a red dot of its middle. A simple recording electrodes are applied on the cornea, forehead and scalp for the electrophysiological measurements. Prior to this procedure a topical anesthetic gel is applied to numb the eye to prevent discomfort from placement of the corneal electrodes.

B. Undergo general eye examination and optical coherence tomography (OCT) to measure the retinal tissue thickness. Prior to eye examination,eye drops are applied into the eyes to enlarge the pupils C. Sit in front of a fundus camera for obtaining images of the retinal vessels to measure oxygen saturation and the vessel width

Researchers will compare the obtained measurements with age- and gender matching of healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Parkinson Disease

Exclusion Criteria:

* Eye disease
* Diabetic Mellitus
* Chronic Obstructive Pulmonary Disease (COPD)
* Other Neurological Disease
* Smoking on a daily basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with confirmed parkinsons disease Stage 0-3 on the Hohen and Yahr scale
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Retinal vessels oxyhemoglobin saturation | Baseline. On the visit to the ambulatory Opthalamic department at Landspitali
  Obtained by retinal oximetry

SECONDARY OUTCOMES:
Vessel width of retinal arterioles and venules | Baseline. On the visit to the ambulatory Opthalamic department at Landspitali
  Obtained by retinal oximetry
Retinal nerve fiber layer thickness | Baseline. On the visit to the ambulatory Opthalamic department at Landspitali
  Obtained by cross-sectional imaging of the retinal tissue (OCT)
Components and waveform of VEPs | Baseline. On the visit to the ambulatory Opthalamic department at Landspitali
  Pattern electroretinogram (PERG)
Pattern electroretinograms (PERGs) | Baseline. On the visit to the ambulatory Opthalamic department at Landspitali
  Amplitude of the visual evoked potential response

CONTACTS AND LOCATIONS:
Overall Officials: Thorunn S Eliasdottir, PhD, CRNA, Principal Investigator — University Hospital of Iceland and University of Iceland. Reykjalundur; Thorunn S Eliasdottir, PhD, CRNA, Principal Investigator — Landpitali the University Hopital of Iceland; Thorunn S Eliasdottir, PhD, CRNA, Principal Investigator — University of Iceland; Soley Thrainsdottir, MD, PhD, Principal Investigator — Reykjalundur
Locations (1):
- Ophthalmic Outpatient Department Landspitali UH, Reykjavik, Iceland